CLINICAL TRIAL: NCT05560750
Title: Lingual Frenulum in Newborn Infants (LINNE): Prospective, Observational Study of the Oral Structural Variations, Their Correlations to the Functional Distinctions, and a Randomized, Controlled Trial on the Treatment of the Tongue-tie
Brief Title: Lingual Frenulum in Newborn Infants (LINNE)
Acronym: LINNE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 83/2022; 2022-001546-37 (EudraCT Number)
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Tongue Tie; Frenulum Breve; Frenulum; Elongation; Breast Feeding
Keywords: Tongue tie; Frenulum lingualis; Frenotomy; Oral physiotherapy; Newborn infant; Breastfeeding; Breastfeeding complications; Logopedic evaluation
MeSH Terms: conditions — Ankyloglossia; Breast Feeding | interventions — Oral Frenectomy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Study patients with parental consent are randomized into 3 study arms:
  1. Open study treatment (index therapy) is a frenotomy performed under local anesthesia or general anesthesia, i.e. an operation to release the lingual frenulum immediately after its detection;
  2. Conservative treatment is a parental given sensitive movement therapy aiming to tongue-tie stretching for 4 weeks;
  3. Follow-up group (no-treatment): appointment for the procedure at one month age with a re-evaluation for the procedure.
Who Masked: Care Provider
Masking Description: One month follow-up time (parents unaware)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Frenotomy (Experimental): Patients who will have frenotomy soon after randomisation, on the same or next day
  Interventions: Procedure: Frenotomy
- Oral physiotherapy (Active Comparator): Patients whose parents are guided to give the child oral physiotherapy for 1 month
  Interventions: Procedure: Oral physiotherapy
- Follow-up (No Intervention): Patients whose frenotomy appointment will be set at 1 month age

INTERVENTIONS:
Procedure: Frenotomy — Releasing the tongue-tie with scissors
  Other Names: Frenulum elongation
  Arms: Frenotomy
Procedure: Oral physiotherapy — Gentle parental activation of the mouth area and the tongue for 1 month
  Arms: Oral physiotherapy

SUMMARY:
Oral cavity's structural variations are involved in the successful breastfeeding of the newborn infants. The tongue-tie has been shown to cause breastfeeding problems. This project investigates the oral structural properties of the newborn infants and the efficacy and safety of their treatment options in breastfeeding problems. The project includes two studies: 1. A prospective follow-up study that investigates the epidemiology and associations between oral structures and breastfeeding problems in term and preterm infants; 2. A randomised, controlled study that investigates the efficacy and safety of tongue-tie treatments. Follow-up visits are planned two to three months, one year, and five years after randomisation along with a 6 months' e-questionnaire for all study patients. The study provides information at the population level.

DETAILED DESCRIPTION:
Part 3 of the LINNE project: Efficacy and safety of neonatal tongue-tie therapies: a controlled, randomised, clinical trial

1 Aim, hypotheses and objectives

Present trial investigates the effectiveness and safety of conservative and surgical treatments of tongue-tie in treatment of neonatal feeding difficulties. The neonatal participants have been diagnosed an anatomical and functional tongue-tie that interferes feeding in the observational study (Project parts 1-2).

Hypotheses

1. A tongue-tie release procedure, frenotomy, indicated by the study tongue-tie criteria, is effective and safe
2. The mother's breastfeeding experience and the parents' satisfaction improve with adequate treatment of the newborn
3. No long-term adverse effects will be detected.

Aims

1. To investigate the efficacy and safety of operative versus conservative treatment of a tongue-tie diagnosed with the study criteria
2. To study the mother's breastfeeding experience and parents' satisfaction to different treatment approaches.
3. To conduct the long-term follow-up of the treatments.

2 Study design

A randomised, controlled, blinded, single-centre, clinical trial. Study arms:

1. Open study treatment (index therapy) is the frenotomy performed under local anaesthesia or general anaesthesia, i.e., an operative release of the tongue-tie immediately after its detection.

   Description of the procedure: During the excision of the tongue-tie, the parent is sitting in a chair with the infant in his/her lap. The child may be lying on the treatment table as well. In both cases, an assistant supports the child's head. Anaesthesia is conducted with medical cream (lidocaine 25 mg/ml and prilocaine 25 mg/ml) that is applied into the floor of the mouth on both sides of the lingual frenulum, up to 1 ml, approximately for 30 sec - 1 min. The anaesthetic then is removed by sweeping by a bandage. The tongue is elevated with a grooved director and the lingual frenulum is cut with scissors to free the tip of the tongue. The release is targeted to the mucosal and connective tissue parts of the lingual frenulum, the muscle fibres will not be cut. It is a quick procedure; 20 minutes will be reserved for the appointment.

   The procedure may result in minor bleeding which can be controlled by compressing it with a bandage moistened with lidocaine-adrenal solution, if necessary. The solution is prepared by mixing 20 ml of Lidocaine 20 mg/ml, and 1 ml of Adrenalin 1 mg/ml. The solution is a generally used topical anaesthetic in otorhinolaryngological (ORL) procedures. Normal bleeding from the procedure usually lasts a few minutes, up to 10 minutes. Due to bleeding, corrective procedures (diathermy) are needed extremely rarely. Afterwards, some bloody stains in the baby pukes are possible and parents will be informed about it.

   As after-care, parent will be guided a physiotherapy of the surgical area to prevent scarring (Annex 3: hospital guidelines). In addition, if necessary, parents are advised to give paracetamol mixture 24mg/ml by the weight-based dosage (15mg/kg) up to three times a day for couple days if the child seems to have pain or discomfort. A control visit takes place one month after the procedure.
2. Conservative treatment includes a sensitive oral physiotherapy aiming to stretch the tongue-tie (Annex 4 and internet video (YouTube)). Treatment will continue up to 4 weeks, unless the Study infant follow-up guideline for urgent treatment criteria, given to the parents at randomisation, would be earlier met (Annex 5). According to the guidelines, the parents may contact investigators any time when necessary. The need for operative treatment is re-evaluated at the follow-up visit after the physiotherapy period, or at an earlier appointment on demand.
3. The follow-up group (no-treatment) receive the appointment date for the procedure at one month after randomisation. However, if the Study infant follow-up guideline criteria (Annex 5) would be met prior to the date given, parents may contact investigators and the appointment would take place earlier.

A two to three minutes video recording of the infants' feeding is documented using the study mobile phone.

The main purpose of the feasibility study is to assess the validity and practicality of the previously unused research components that are essential and unique to the present trial. These include e.g. the study anatomical-functional scoring, oral physiotherapy, and the blinding method of the parents. According to the preliminary plan, the trial will be conducted using the same formulations as the feasibility pilot, but some details of the final design, as well as the sample size estimation, will be checked upon the feasibility study results.

3 Sample size

Feasibility study:

According to a previous study, the harm caused by a tongue-tie had been disappeared in 92% of the operated children three months after the procedure. In the group of non-operated control patients, 47% reported that the harm disappeared without the procedure. According to the null hypothesis of this feasibility study, the groups do not differ, i.e., the treatments have no effect on breastfeeding success. With 80% power and 5% alpha error, the required sample size is 15 infants/group. Due to the randomisation to three groups, n=48 is needed, resulting in a group size of n=16.

Randomised clinical trial (RCT):

In a previous six-year follow-up study of Dept. of Otorhinolaryngology, Oulu University Hospital (2013-2018), 365 tongue-tie diagnoses were done, mean 61/year. The number of operative treatments was 334, i.e., 56/year. For the final sample size calculation, the change in the primary outcome required will be checked upon the feasibility pilot. An educated guess is approximately 300 infants (100/group).

4 Blinding and randomization

The study physician will discuss with the parents and request the written informed consent.

An assigned randomisation executor, beyond the study group, will conduct the computed randomisation of the trial code numbers prior to the beginning of the trial. The codes will be written upon the opaque envelopes, containing information of the study therapy group in question.

After the informed consent, the infant will be assigned the next free trial code from the list. The investigator opens the envelope marked by the code number, in which the treatment group information is placed. The study nurse organizes the follow-up visits and guides with the treatment and follow-up instructions.

5 Follow-up protocols

Patients will be invited to an evaluation visit by a speech therapist at the age of 2-3 months. The research will be carried out at Oulu University Hospital. A speech therapist, specialising in neonatal feeding, will be blinded to the patient's treatment group. Infant sucking pattern, interruptions in sucking, irritability during breastfeeding, possible flatulence, and possible breastfeeding problems are evaluated.

The trial patients are invited to outpatient clinic control visits at the age of 1 and 5 years.

At the age of one year (12 ± 2 mo) control visits, eating patterns (sucking, swallowing, biting, chewing, drooling, eating solid foods, cleaning the mouth by tongue, resting position of the tongue, licking, sweeping around the lips by the tongue), presence of mouth breathing, and dentition development are assessed. The examination may be videotaped, and if necessary, with a separate parental permission, specifically if the child has an eating or speech defect. Control visits take place at the Oulu University Hospital ORL-department by study physicians.

At the age of five years (exclusion criteria: diagnoses affecting speech and language development), the production of sounds requiring tongue tip raising ([t, d, n, l, s, r], including a total of 30 words, 5 per sound) is assessed by the child naming them from pictures. Should the naming be not successful, the child will be asked to repeat. The discussion will take only a short time, or the child will be asked to tell. The visit will be videotaped. A logopedic assessment group will evaluate the abnormalities of articulation (abnormal/not) and intelligibility of the speech (VAS scale), and by using a four-point Likert scale whether the possible articulation errors affect the intelligibility of the speech. In addition, the parents will be asked about the child's eating habits and possible problems.

6 Data management

Patient data as well as study videotapes will be recorded to the electronic research database, the study hospital's M-drive, that can be accessed only by study team members. The data of the children participating in the trial is collected from the study files and e-mail questionnaires. Information necessary for the study is stored in the database. All paper documents are kept in the closed office of the principal investigator until the official storage period of the research archive has ended. A self-assessment of the security risks of the study data has been stated for parental access upon demand.

Only the study personnel know the identity and other identifiable information of the study patients, and they are all bounded by secrecy. All data are processed and coded in such a way that individual information cannot be identified from the study results. An inspector external to the study (monitor) has the right to revise the study documents if necessary.

7 Statistical methods

Special statistical program (IBM SPSS) will be used for statistical analyses. Continuous variables will be analysed with a t-test or non-parametric tests, depending on the distribution. Chi2 or Fisher's exact tests are used for the analysis of dichotomous variables. Analyses of associations are performed with Pearson's, Spearman's or Kendall's correlation coefficients and, if necessary, variance or regression analyses (Risk ratio, Odds ratio, numbers needed to treat). Consistency between researchers is tested with the Kappa coefficient. The results will be analysed according to the intention-to-treat principle. The limit of statistical significance is set at p<0.05.

8 Study permits and practices

The trial authorization of the regional ethics committee has been applied and permitted. Permission for the clinical study is being sought from the administrative management of Oulu University Hospital.

The research will be conducted the principles of Good Clinical Practice (GCP). An external monitor will be appointed for the study for the implementation of the study and the fulfilment of the patients' rights.

The hospital patient insurance covers all the study patients. Patients will not be compensated for participating in the trial, with the exception of normal parental accompanying costs.

9 Quality and appropriateness of the premises and equipment of the trial sites

The Oulu University Hospital's Mother-Child Unit, Department of Otorhinolaryngology, Neonatal Intensive Care Unit, Neonatal ward, and Faculty of Humanities, Research Unit of Logopedics, are the study sites. The qualifications of the personnel of these units are appropriate for the implementation of the research. The equipment of the tertiary-level hospital and the emergency facilities are modern and appropriate for study safety.

10 Timetable estimation

Prospective study will be launched during the fall of 2022. The recruitment will last for an estimated three years, and the follow-up protocol will continue for another five years. The first analyses and reporting of the results of the feasibility study will be done during 2023-2024.

11 Funding

The present project will be carried out using personal and project grants, applied from the medical research foundations. The study represents an investigator-driven research and will be executed without commercial funding. The project has no connections to the pharmaceutical or any other commercial companies.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infant with at tongue-tie interfering the breastfeeding and patient's study screening scoring exceeding >8/19

Exclusion Criteria:

* Child's severe anomaly or illness; the parent's severe illness; a communication problem between parents and researchers (e.g. language barrier); any other practical reason that prevents the child to have the procedure or the parents to provide the oral physiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful breastfeeding | 1 month age
  Mother breastfeeding the child w/o problems

SECONDARY OUTCOMES:
Anatomical classification of the frenulum lingualis | 1 month
  TABBY scoring
Histological classification of the frenulum lingualis | 1 month
  Classification a.m. Mills et al
Height of the oral cavity | 1 month
  Measurement from the hard palate to the upper alveolar crest, cm
Width of the jaw | 1 month
  Interramal measurement, cm
Breastfeeding problems questionnaire | 1 month
  Symptoms of the mother or the infant
Breastfeeding problems' reasons | 1 month
  Any reason for prohibiting/complicating the breastfeeding
Duration of breastfeeding | 6 months
  Duration of total and partly breastfeeding, weeks
Daily crying time of the infant | 24 h
  Parents' approximation of how long time the infant cries during a day, hours
Infant's morbidities | 6 months
  The diagnoses made by doctors
Infant's weight growth | 1 year
  Weight, kg
Infant's height growth | 1 year
  Height, cm
Infant's head growth | 1 year
  Head circumference, cm
Maternal breastfeeding experience, questionnaire | 6 months
  Subjective evaluation
Parents' satisfaction, questionnaire | 6 months
  Subjective evaluation
Complications of the possible procedures | 1 month
  Frenotomy or physiotherapy complications diagnosed by physicians

OTHER OUTCOMES:
Speech therapy evaluations and their results | 5 years
  Logopedic evaluations' results

CONTACTS AND LOCATIONS:
Overall Officials: Outi Aikio, MD, PhD, Principal Investigator — Oulu University Hospital, Dept of Pediatrics; PEDEGO Research unit and MRC Oulu, University of Oulu
Locations (3):
- Finland (3):
  - Department of Otorhinolaryngology, Oulu University Hospital, Oulu
  - Department of Pediatrics, Oulu University Hospital, Oulu
  - University of Oulu, Faculty of Humanities, Research Unit of Logopedics, Oulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A review article on the treatment of the tongue tie — https://www.laakarilehti.fi/tieteessa/katsausartikkeli/kirea-kielijanne-ja-hammentava-huulijanne-ndash-pitaako-hoitaa/